CLINICAL TRIAL: NCT02999334
Title: HIV With Innovative Group Antenatal Care in Two African Countries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Crystal L. Patil, PhD, Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NR14413-01
Record Dates: First submitted 2016-12-11; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Prenatal Care
Keywords: Group healthcare models; Antenatal care; Prenatal care; Perinatal health; CenteringPregnancy; sub-Saharan Africa; Malawi; Tanzania; Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Individual ANC (standard care) (No Intervention): Individual ANC is the standard of care. Women arrive at the clinic and and are provided ANC services on a first come, first serve basis. While waiting women who are present listen to a health lecture. Women then complete laboratory tests, including HIV testing (at the first visit), then meet individually with a midwife for a brief one-on-one physical assessment. Four ANC visits are recommended.
- Group ANC (intervention) (Experimental): Women in CP-based group antenatal care (intervention) arrive at clinic at the scheduled appointment time and go directly to the group space. The same group of 12 women and the midwife and co-facilitator are present at each session. Women measure and record their own vital signs and weight. Each then has a brief one-on-one assessment with the midwife in the group space room. Instead of health lectures, the group engages in facilitated and interactive discussions using activities. Four ANC visits are recommended.
  Interventions: Behavioral: Group Antenatal Care

INTERVENTIONS:
Behavioral: Group Antenatal Care — To examine the effect of type of care on completion of the recommended antenatal and postnatal visits as well as perinatal health outcomes, including knowledge, behaviors, psychosocial well-being, pregnancy-related empowerment, satisfaction with ANC care.
  Arms: Group ANC (intervention)

SUMMARY:
The quality of antenatal care (ANC) in much of sub-Saharan Africa is constrained by severe resource and staffing shortages. The investigators adapted and piloted an evidence-based model of group antenatal care as an innovative way to improve ANC service delivery and increase health promotion. This pilot will be conducted in Malawi and Tanzania and will provide data to prepare for a large randomized controlled trial to document the impacts that group antenatal has on perinatal health outcomes. This study will ultimately inform policy and practice aimed at improving quality of antenatal care through respectful and woman-centered care to pregnant women.

DETAILED DESCRIPTION:
More than 90% of women in sub-Saharan Africa use antenatal care (ANC) at least once in pregnancy. To leverage high attendance rates, most facilities bundle HIV prevention and prevention of maternal-to-child transmission (PMTCT) with ANC. Unfortunately, the quality of ANC in sub-Saharan Africa is sharply constrained by severe resource and staffing shortages, as reflected in numerous "missed opportunities" for PMTCT, clinical service delivery, and health education. Moreover, job satisfaction among the overburdened providers is low. To improve ANC quality, the investigators will adapt and pilot an innovative, evidence-based model of group ANC, an approach that restructures provider time, allowing health facilities to offer respectful, woman-centered and high quality ANC given the limitations.

In CenteringPregnancy (CP), the only evidence-based model of group ANC, 12 women meet jointly for two hour antenatal visits, assessing their own weights and blood pressures, meeting briefly with the provider for individual consultations, and engaging in facilitated health discussions. Randomized controlled trial (RCT) data from ethnically and socioeconomically diverse populations in the US demonstrated that CP is highly effective at improving ANC adherence, provider and client satisfaction, and maternal and child outcomes. In the US, the successful integration of HIV prevention into the CP model reduced sexually transmitted infections and increased condom use.

CP has not been implemented with fidelity and tested for efficacy in a low-resource country. With funding from the Chicago Developmental Center for AIDS Research, the investigators conducted preliminary work in Malawi and Tanzania which suggested that a CP-based model of group ANC was feasible and acceptable; both women and providers were excited and energized by the model. The purpose of this study is to build on this work and: 1) conduct the developmental work to collaboratively adapt CP materials for use in both countries (sessions, training guides, and implementation and evaluation strategies); 2) train providers and pretest activities; and 3) conduct a full-scale randomized pilot. Investigators will work directly with the Centering Healthcare Institute to implement this CP-based model of group ANC with fidelity. This study will result in a feasible, acceptable, and sustainable CP-based model of group ANC adapted for the constraints posed by poorly resourced health systems and those of the clients they serve. These pilot data will be used to generate retention rates and effect sizes for an RCT to test the efficacy of a CP-based group ANC model.

Group antenatal care is an innovative paradigm shift in ANC, and this rigorous evaluation of its impact will expand the limited scientific assessments of reconfigured ANC models and mother and infant health outcomes in low-resource countries in sub-Saharan Africa. Because this model was developed and tested in target countries with high HIV prevalence and poor maternal and neonatal outcomes, it has the potential for broad impacts on maternal and child health, including PMTCT, in other low resource settings.

ELIGIBILITY:
Inclusion Criteria:

* Physically and mentally competent pregnant women over the age of 16 attending antenatal care

Exclusion Criteria:

* Less than 16 years of age

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2013-09; Primary Completion 2015-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Adherence to Care | 6-8 weeks postpartum
  Two Indicators: Attended 4 (or more) antenatal care visits (yes, no) and the 6-week postnatal visit (yes, no)

SECONDARY OUTCOMES:
Healthy Pregnancy Knowledge Index | Enrollment, 32-40 weeks gestation
  14-item true/false questions measured two times in pregnancy and scored as percent correct (range 0-100%)
Healthy Pregnancy Behaviors | Enrollment, 32-40 weeks gestation
  Substance use behaviors in the last two months for: tobacco products, alcohol, and marijuana. Two nutritional behaviors were asked about. One was whether or not she ate fruits or vegetables at least 3 times a day for 5 or more days in the past week. The second focused on eating protein at least once a day for 5 or more days in the past week. Measured two times in pregnancy. Three or less of these five behaviors scored as 0 and four or more healthy behaviors were categorized as a 1 (Dichotomous)
Prevention of Mother-to-Child (PMTCT) Knowledge | Enrollment, 32-40 weeks gestation
  4-item PMTCT knowledge index measured two times in pregnancy and scored as 1 if all four were correct and 0 if one or more item was incorrect (Dichotomous)
Comprehensive HIV Prevention Knowledge | Enrollment, 32-40 weeks gestation
  5-item comprehensive HIV knowledge index measured twice in pregnancy. Scored as 1 if all five items were correctly and 0 if one or more item was incorrect (Dichotomous)
Mental Distress | Enrollment, 32-40 weeks gestation
  20-item yes/no Self Reporting Questionnaire (SRQ-20) to assess mental distress was measured two times in pregnancy. Validated in multiple countries including Malawi and Tanzania (Range 0-20, baseline α = 0.789; late pregnancy α = 0.848). We dichotomized scores to low (<8 symptoms) and high (≥8), a level used in clinics for referral. (Dichotomous)
Pregnancy-Related Empowerment Scale (PRES) | 32-40 weeks gestation
  The pregnancy-related empowerment scale (PRES) is a 16-item Likert-type scale with items ranging from 1 (strongly disagree) to 4 (strongly agree) that is intended to assess a woman's sense of control over their pregnancy health and health care. Measured once in late pregnancy (Range 16-64, Continuous)
Satisfaction with Care | 32-40 weeks gestation
  10-item satisfaction with antenatal care index; Measured once in late pregnancy with 5 response options between 1 (poor) and to 5 (excellent) (Range 13-50, Continuous)
Any Adverse Perinatal Event | 6-8 weeks postpartum
  Fetal demise, stillbirth, neonatal death, preterm birth, low birth weight, or maternal death. None experienced = 0; one or more = 1 (Dichotomous)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal L Patil, PhD, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patil CL, Abrams ET, Klima C, Kaponda CP, Leshabari SC, Vonderheid SC, Kamanga M, Norr KF. CenteringPregnancy-Africa: a pilot of group antenatal care to address Millennium Development Goals. Midwifery. 2013 Oct;29(10):1190-8. doi: 10.1016/j.midw.2013.05.008. Epub 2013 Jul 19. PMID 23871278
- [Derived] Liese KL, Kapito E, Chirwa E, Liu L, Mei X, Norr KF, Patil CL. Impact of group prenatal care on key prenatal services and educational topics in Malawi and Tanzania. Int J Gynaecol Obstet. 2021 Apr;153(1):154-159. doi: 10.1002/ijgo.13432. Epub 2020 Dec 2. PMID 33098114
- [Derived] Patil CL, Klima CS, Steffen AD, Leshabari SC, Pauls H, Norr KF. Implementation challenges and outcomes of a randomized controlled pilot study of a group prenatal care model in Malawi and Tanzania. Int J Gynaecol Obstet. 2017 Dec;139(3):290-296. doi: 10.1002/ijgo.12324. Epub 2017 Oct 10. PMID 28905377